CLINICAL TRIAL: NCT05354128
Title: Intravenous Thrombolysis Versus Primary PCI for Recanalization Time in Acute ST-segment Elevation Myocardial Infarction in the Context of the COVID-19 Outbreak: a Prospective, Multicenter, Nonrandomized Controlled Registry Study.
Brief Title: Thrombolysis in STEMI Patients Compared With pPCI on Recanalization Time in the Context of the COVID-19 Outbreak.
Acronym: RESCUE-STEMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ya-Wei Xu (Other)
Responsible Party: Sponsor-Investigator, Ya-Wei Xu, Director of the Heart Center, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESCUE-STEMI
Record Dates: First submitted 2022-04-27; First posted 2022-04-29 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Fibrinolytic Agents

STUDY DESIGN:
Intervention Model Description: non-randomized control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrombolysis Group (Experimental): Patients who meet the conditions for intravenous thrombolysis are included in the intravenous thrombolysis group. Regardless of whether the thrombolysis is successful or not, CAG examination is performed afterwards to clarify the vascular condition, and PCI is performed if necessary.
  Interventions: Drug: Thrombolytic
- PCI Group (Other): Eligible patients undergoing primary PCI.
  Interventions: Procedure: percutaneous coronary stenting

INTERVENTIONS:
Drug: Thrombolytic — Standard intravenous thrombolysis.
  Other Names: intravenous thrombolysis
  Arms: Thrombolysis Group
Procedure: percutaneous coronary stenting — Percutaneous coronary stenting
  Other Names: PCI
  Arms: PCI Group

SUMMARY:
During the outbreak of COVID-19, for patients with acute ST-segment elevation myocardial infarction with unclear infection, the time of primary PCI is uncertain, and it is often expected to exceed 90 minutes or even 120 minutes. In indicated patients, intravenous thrombolysis has significantly improved the recanalization time of criminal vessels.

DETAILED DESCRIPTION:
During the outbreak of COVID-19, for patients with acute ST-segment elevation myocardial infarction with unclear infection, the time of primary PCI is uncertain, and it is often expected to exceed 90 minutes or even 120 minutes. In indicated patients, intravenous thrombolysis has significantly improved the recanalization time of criminal vessels. The purpose of this study was to compare the time from first medical contact to patency and safety (specifically symptom improvement, ECG ST segment) between intravenous thrombolysis and concurrent patients with possible primary PCI in a prospective, multicenter, non-randomized controlled manner. Significant fall, angiographic examination showed criminal blood vessel TIMI blood flow grade 2-3)

ELIGIBILITY:
Inclusion Criteria:

* ECG confirms acute ST-segment elevation myocardial infarction；The estimated time from FMC to recanalization is more than 120 minutes；

Exclusion Criteria:

* Intracranial hemorrhage or stroke within the past 6 months; central nervous system injury, tumor or arteriovenous malformation; bleeding disease with known cause; suspected aortic dissection; non-compressible puncture surgery within 24 hours, etc.; 1 week of pregnancy or postpartum; uncontrolled hypertension; advanced liver disease; active peptic ulcer; prolonged or invasive CPR;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
recanalization | within 24 hours
  Coronary angiography to check for recanalization after thrombolysis（Yes or No）
recanalization time | within 2 hours
  From first medical contact(FMC) time to recanalization time.

SECONDARY OUTCOMES:
Major bleeding event | 7 day
  Whether there is a major bleeding event with drug thrombolysis（Yes or No）
Malignant arrhythmia | 12 hours
  Malignant arrhythmia incidence

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, Doctor, Study Director — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No